CLINICAL TRIAL: NCT07020091
Title: Predictors of In-Hospital Mortality in Patients With Return of Spontaneous Circulation After Cardiac Arrest: A Prospective Observational Study
Brief Title: Predicting Mortality in Patients With Return of Spontaneous Circulation After Cardiac Arrest
Acronym: PROM-ROSC
Status: Active, not recruiting | Type: Observational
Sponsor: Ahmet Düzgün (Other)
Responsible Party: Sponsor-Investigator, Ahmet Düzgün, Specialist in Internal Medicine and Intensive Care, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Organization: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Other Study IDs: GAZI-494-ROSC-2025; GAZI-ROSC-494-2025 (Other: Gazi Yaşargil Training and Research Hospital Ethics Committee)
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Post-Resuscitation Syndrome; Critical Illness; Cardiac Arrest; Hypoxic-Ischemic Encephalopathy; Coma
Keywords: Cardiac Arrest; ROSC; In-Hospital Mortality; ICU; Post-Resuscitation Care; Neurological Outcome
MeSH Terms: conditions — Critical Illness; Heart Arrest; Hypoxia-Ischemia, Brain; Coma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ROSC Cohort: Adult patients (≥18 years old) who achieved return of spontaneous circulation (ROSC) after cardiac arrest and were admitted to the intensive care unit. These patients are prospectively followed to evaluate clinical and biochemical predictors of in-hospital mortality.

SUMMARY:
This observational study aims to identify early predictors of in-hospital mortality in adult patients who achieved return of spontaneous circulation (ROSC) after cardiac arrest. The study prospectively enrolls patients admitted to the intensive care unit at a tertiary care hospital in Turkey. Various clinical, biochemical, and resuscitation-related parameters will be recorded within the first 24 hours of ICU admission. The primary goal is to determine which factors are most strongly associated with mortality within 30 days. The findings are expected to improve clinical decision-making and risk stratification in the management of post-cardiac arrest patients.

DETAILED DESCRIPTION:
This is a prospective observational study conducted in the intensive care unit (ICU) of Gazi Yaşargil Training and Research Hospital, Turkey. The study aims to identify independent predictors of in-hospital mortality in patients who achieve return of spontaneous circulation (ROSC) after cardiac arrest. Adult patients (age ≥ 18 years) who were resuscitated after cardiac arrest and admitted to the ICU are consecutively included.

Data are collected prospectively on admission and within the first 24 hours, including demographic characteristics, cause and type of arrest, time to ROSC, initial rhythm, hemodynamic parameters, neurological status, lactate, pH, base excess, biomarkers, and therapeutic interventions. Primary outcome is 30-day in-hospital mortality. Secondary outcomes include neurological outcome at discharge and ICU length of stay.

Patients are followed up until hospital discharge or death. The data will be analyzed using multivariate logistic regression to identify independent risk factors for mortality. The study was approved by the institutional ethics committee, and no intervention beyond routine care is performed. Results are expected to improve clinical prognostication and guide decision-making for patients with ROSC after cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Achieved return of spontaneous circulation (ROSC) after cardiac arrest
* Admitted to the intensive care unit (ICU)
* Informed consent obtained from patient or legal representative (if applicable)

Exclusion Criteria:

* Age < 18 years
* Known pregnancy
* Brain death at the time of ICU admission
* Patients with missing key clinical or laboratory data
* Declined participation or legal refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years old) who achieved return of spontaneous circulation (ROSC) after cardiac arrest and were admitted to the intensive care unit (ICU) at Gazi Yaşargil Training and Research Hospital, Turkey. Patients are consecutively enrolled and observed for outcomes related to in-hospital and 6-month mortality.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
In-Hospital Mortality | From ICU admission to hospital discharge (up to 60 days)
  All-cause mortality recorded during the index hospital stay following return of spontaneous circulation (ROSC).
6-Month Mortality | 6 months after ICU admission
  All-cause mortality assessed at 6 months following the initial cardiac arrest event. Mortality status is confirmed through hospital records and national death registry.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi Yaşargil Training and Research Hospital, Diyarbakır, kayapinar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
At this stage, no final decision has been made regarding individual participant data (IPD) sharing. The possibility of sharing anonymized IPD will be evaluated after the study is completed and initial results are published, taking into account ethical, legal, and institutional considerations.